CLINICAL TRIAL: NCT01481493
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Dose-finding Study in Patients With Active Rheumatoid Arthritis Incompletely Controlled on Stable MTX Doses to Investigate Efficacy and Safety of SC BT061
Brief Title: Dose-finding of Multiple Dose of BT061 in Patients With Active Rheumatoid Arthritis Incompletely Controlled on Stable Methotrexate (MTX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 979; 2010-018485-24 (EudraCT Number)
Record Dates: First submitted 2011-10-17; First posted 2011-11-29 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Experimental): BT061 monoclonal antibody (subcutaneous)
  Interventions: Biological: BT061
- Placebo (Placebo Comparator): subcutaneous injection of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BT061 — subcutaneous administration of the monoclonal antibody BT061
  Other Names: immune-modulatory antibody BT061
  Arms: Active Treatment
Biological: Placebo — subcutaneous injection of placebo
  Other Names: end formulation buffer without active ingredient
  Arms: Placebo

SUMMARY:
The study is conducted in order to find out if repeated doses of the monoclonal (artificially manufactured) antibody BT061 can help arthritis patients whose disease does not sufficiently respond to a treatment with methotrexate (MTX).

DETAILED DESCRIPTION:
Patients showing active rheumatoid arthritis according to ACR criteria despite at least 6 months of treatment with methotrexate fulfilling all other inclusion criteria including written informed consent and none of the exclusion criteria (see below) have the opportunity to be randomised to either treatment with BT061 or placebo, both given subcutaneously in a double-blind set-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Rheumatoid Arthritis (RA) according to 1987 revised ACR criteria with functional class II-III
* Disease activity at screening and baseline (more than 6 swollen joint count; more than 6 tender joint count; elevat. of CRP or ESR)
* Duration of RA more than 12 month
* History of at least one disease-modifying anti-rheumatic drug (DMARD) with an inadequate response despite more than 3 month of treatment
* MTX treatment at least 6 month with a stable dose at least 15mg MTX
* Patients could continue at more than daily 7,5mg of prednisone or equivalent stable dose at least 6 weeks prior baseline
* Written Informed Consent

Exclusion Criteria:

* Treatment with traditional DMARDs apart from MTX 12 weeks prior to baseline and DMARD leflunomide 24 weeks
* Treatment with any biologics other than TNF-α inhibitors (e.g. abatacept, rituximab, tocilizumab, anakinra)
* treatment with any TNF-α inhibitor within 5 elimination half-lives prior baseline and during the study
* Clinical non-response to more than one of TNF-α inhibitor exceeding adequate treatment duration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
dose-response information | ACR20 response at week 13 (1 week after last dose of study drug)
  ACR20 response (percentage of patients reaching or exceeding at least a 20% improvement in their arthritis assessment according to the criteria of the American College of Rheumatology)

SECONDARY OUTCOMES:
efficacy responses other than ACR20, including questionaires, and their dose dependencies | weekly assessment of ACR arthritis status during the 12 weeks' treatment course, then repeatedly within 1 to12 weeks after the last dose of study drug
  ACR50, ACR70, ESR, DAS28, CRP, HAQs, FACIT, RF, Hb,
Safety and tolerability of the various dose levels and of placebo | weekly assessment of physical status, safety labs, adverse events during the 12 weeks' treatment course, then repeatedly within 1 to12 weeks after the last dose of study drug
  Physical examinations Vital Signs, Safety Lab, assessment of adverse events, tolerability
Pharmakokinetics (PK) | weekly blood sampling during the 12 weeks' treatment course, then repeatedly within 1 to12 weeks after the last dose of study drug
  BT061 plasma levels, AUC, time to elimination, accumulation after multiple doses, time course of related hematological parameters (e.g. WBC count)

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Vencovský, MD, Study Chair — Institute of Rheumatology, Na Slupi 4, 128 50 Praha 2, Czech Republic
Locations (39):
- Czechia (4):
  - Study Site, Ostrava
  - Study Site, Prague
  - Study Site, Uherské Hradiste
  - Study Site, Zlín
- Germany (5):
  - Study Site (Berlin 1), Berlin
  - Study Site (Berlin 2), Berlin
  - Study Site, Erlangen
  - Study Site, Frankfurt
  - Study site, München
- Hungary (2):
  - Study Site, Nyíregyháza
  - Study Site, Székesfehérvár
- Italy (8):
  - Study Site, Bari
  - Study Site, Cagliari
  - Study Site, Chieti
  - Study Site, Florence
  - Study Site, Genova
  - Study site, Milan
  - Study site, Padua
  - Study Site, Palermo
- Latvia (2):
  - Study site, Daugavpils
  - Study site, Riga
- Poland (11):
  - Study Site (Bialystok 2), Bialystok
  - Study Site, Bialystok
  - Study Site, Bydgoszcz
  - Study Site, Elblag
  - Study site, Gmina Końskie
  - Study Site, Krakow
  - Study Site, Lublin
  - Study Site, Poznan
  - Study Site, Torun
  - Study site, Warsaw
  - Study Site, Wroclaw
- Spain (7):
  - Study site (Barcelona 1), Barcelona
  - Study site (Barcelona 2), Barcelona
  - Study Site, Bilbao
  - Study Site (Madrid2), Madrid
  - Study Site, Madrid
  - Study Site, Málaga
  - Study Site, Santander